CLINICAL TRIAL: NCT00083733
Title: Procurement of Normal Breast Tissue and Metastatic Breast Cancer Tissue for Molecular Profiling
Brief Title: Genetic and Protein Profiling in Normal and Cancerous Breast Tissue
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040199; 04-C-0199; NCT00899938 (obsolete NCT alias)
Record Dates: First submitted 2004-05-29; First posted 2004-05-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-17

CONDITIONS: Breast Neoplasms
Keywords: Gene Expression; Microarray; Stem Cell; Proteomics; Metastases; Breast Tissue; Normal Breast Tissue; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

SUMMARY:
This study will collect, analyze, and compare genes and proteins in normal breast tissue with those in various tissues from women with breast cancer to look for changes that are unique to breast cancer cells. Information about these differences may lead to more effective breast cancer treatments with fewer side effects. The study has the following objectives:

* To define the molecular (genetic and protein) profile of normal breast tissue from pre- and post-menopausal women of different ages and who have had varying numbers of children (or no children), and who are in different phases of the menstrual cycle
* To define the molecular profile of primary breast tumors and tumors that have metastasized (spread) beyond the primary site
* To characterize breast cancer stem cells and establish cell lines from the pleural fluid (fluid around the lungs) of women with metastatic breast cancer. (A cell line is a collection of cells that are grown in the laboratory from an original tissue specimen.)

The following women may be eligible for this study:

* Women who are undergoing cosmetic breast surgery that requires removal of some breast tissue (e.g., breast reduction surgery)
* Women 18 years of age or older who are undergoing a biopsy or other surgical procedure to sample or remove a known or suspected primary or metastatic breast tumor
* Women 18 years of age or older who are undergoing pleurocentesis, a procedure to remove fluid from around the lung that is suspected or known to be caused by spread of breast cancer

Participants undergo the required procedure (e.g., surgery, biopsy, or pleurocentesis) and provide information that may include the following:

* Age, race/ethnicity
* Age at first menstrual period (menarche)
* Age at first pregnancy and age when the first child was born
* Age at menopause
* Information about primary breast cancer
* Family history of breast cancer
* Information on previous breast biopsies, if any, and hormones taken (birth control pills or hormone replacement therapy), if any
* Copy of pathology report from procedure (surgery, biopsy, or pleurocentesis)

DETAILED DESCRIPTION:
Background: Defining the molecular profile (gene and protein expression) of normal breast tissue is essential to identifying markers for cellular subtypes in the normal human breast. These markers could serve as biomarkers for prevention trials or represent new therapeutic targets if they are also expressed in early breast cancers. The gene and protein expression in normal breast tissue may be dependent on the stage of the menstrual cycle, whether the woman is pre- or post-menopausal, prior pregnancy and breast feeding history, and age. The molecular profile of metastatic breast tumors may differ from that of the primary tumor and differ in metastases from different anatomic sites. Identification of genes/proteins unique to these lesions may help identify the processes responsible for metastatic spread at a molecular level and lead to the development of new molecularly targeted drugs. Similarly, isolation and characterization of breast cancer stem cells could provide new approaches for the treatment and prevention of breast cancer.

Objectives: To define the molecular profile of normal breast tissue from pre- and post-menopausal women of varying age and parity (nulliparous to multiparous) and in different phases of the menstrual cycle; to study the molecular profile of primary and metastatic breast cancer lesions; and to identify and characterize breast cancer stem cells and establish cell lines from the pleural fluid of women with breast cancer and malignant pleural effusions.

Eligibility: Women who are undergoing cosmetic breast surgery that entails resection of a portion of the breast (e.g., reduction mammoplasty) and who do not have a history of breast cancer; women with known or suspected breast cancer who are having a primary tumor biopsied or resected or having a metastatic lesion biopsied or resected; or women with breast cancer who are undergoing pleurocentesis for a suspected or known malignant pleural effusion.

Design: Normal breast tissues from cosmetic breast procedures that are performed in women without a history of breast cancer at Suburban Hospital will be snap frozen in liquid nitrogen and sent to the NCI for storage and analysis. Demographic information will be collected from the women undergoing the procedure. Similarly, a portion of biopsies obtained from primary or metastatic lesions in women with suspected or known breast cancer at Suburban Hospital or the NIH will be collected after materials are obtained for diagnostic purposes, snap frozen in liquid nitrogen, and sent to the NCI with demographic information. The unneeded fluid from pleurocenteses performed in women with breast cancer and malignant pleural effusions will be transported (unfrozen) to an NCI lab for immediate processing (FAC sorting to isolate breast cancer stem cells). RNA will be extracted from tissues and cDNA microarrays will be used to study gene expression. Proteomic analysis of normal and malignant breast tissue will be studied using reverse-phase tissue lysates.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects of any age who are undergoing cosmetic breast surgery that entails resection of breast tissue (e.g., reduction mammoplasty) for any reason.
  2. Women (18 years of age or older) with known or suspected breast cancer who are undergoing a diagnostic biopsy or resection of a primary breast lesions or a site of metastatic tumor.
  3. Women (18 years of age or older) with breast cancer who are undergoing a pleurocentesis for removal of fluid from a known or suspected malignant pleural effusion.
  4. All patients or their legal guardians (if the patient is less than 18 years of age) must sign a document of informed consent indicating their understanding that the specimens collected and demographic information provided is only for research purposes. Written assent will be obtained from pediatric patients (less than 18 years of age).

EXCLUSION CRITERIA:

1. Subjects who are undergoing cosmetic breast procedures such as reduction mammoplasty (collection of normal breast tissue) are excluded if they have a prior history of breast cancer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2004-05-27; Study Completion 2010-11-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Russo J, Rivera R, Russo IH. Influence of age and parity on the development of the human breast. Breast Cancer Res Treat. 1992;23(3):211-8. doi: 10.1007/BF01833517. PMID 1463860
- [Background] Russo J, Ao X, Grill C, Russo IH. Pattern of distribution of cells positive for estrogen receptor alpha and progesterone receptor in relation to proliferating cells in the mammary gland. Breast Cancer Res Treat. 1999 Feb;53(3):217-27. doi: 10.1023/a:1006186719322. PMID 10369068
- [Background] Hovey RC, Trott JF, Vonderhaar BK. Establishing a framework for the functional mammary gland: from endocrinology to morphology. J Mammary Gland Biol Neoplasia. 2002 Jan;7(1):17-38. doi: 10.1023/a:1015766322258. PMID 12160083